CLINICAL TRIAL: NCT04042090
Title: A Pilot Study on the Efficacy, Acceptability, Tolerability and Feasibility of a Therapeutic Virtual Reality Application on Improving the Quality of Life in Non-specific Chronic Low-back Pain Patients
Brief Title: The Efficacy, Acceptability, Tolerability and Feasibility of a Therapeutic Virtual Reality Application
Acronym: PijnVRij
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL70042.091.19; 2019-5441 (Registry Identifier: CMO); 2019-5441 (Other: Radboudumc valorisation)
Record Dates: First submitted 2019-07-05; First posted 2019-08-01 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2020-07

CONDITIONS: Back Pain Lower Back Chronic; Quality of Life
Keywords: Virtual reality; Quality of life; Back pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned (1:1) to either the intervention group or the control group. Both intervention and control group are placed on the waiting list (approximate time of waiting is 6 weeks) to receive treatment. Meanwhile, our study will be executed. Intervention group: use of virtual reality intervention at home over a period of 28 days (with a maximum of 35 days) at least ten minutes a day (excluding day 1, in which the participants should do the entire education module of 25 minutes) and in addition, when participants feel the need. The control group: no intervention, patient is waiting to receive normal chronic pain treatment. Randomisation is not blinded: both researchers and participants know which participants are part of the intervention and control group. Randomisation will take place using a computerised randomisation list with variably sized blocks, directly after providing oral informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: use of therapeutic virtual reality (Experimental): Intervention group: use of virtual reality intervention at home over a period of 28 days (with a maximum of 35 days) at least ten minutes a day (excluding day 1, in which the participants should do the entire education module of 25 minutes) and in addition, when participants feel the need. Meanwhile, participant is placed on the waiting list to receive normal chronic pain treatment.
  Interventions: Device: Reducept, virtual reality
- Control group: no use of therapeutic virtual reality (No Intervention): Control group: no intervention, patient is waiting to receive normal chronic pain treatment.

INTERVENTIONS:
Device: Reducept, virtual reality — The VR serious game Reducept is a novel psychological VR intervention for treating chronic pain. It incorporates several psychological therapies into one application: hypnotherapy, mindfulness, ACT and EMDR. Reducept has been made in co-creation with patients, researchers, psychologists and developers and can be installed and played on a VR goggles. It consists of an education module and three games.
  Arms: Intervention group: use of therapeutic virtual reality

SUMMARY:
This study evaluates the effect of therapeutic Virtual Reality (VR) on quality of life of 60 patients with non-specific chronic low-back pain. 30 patients will be included in the intervention group. These patients will use Reducept, a therapeutic virtual reality application based on diverse cognitive therapies (ACT, mindfulness, EMDR, hypnotherapy), at home over a period of 28 days, for at least 10 minutes each day. This will be an add-on intervention next to standard care, while the patient is waiting to receive actual treatment for chronic pain. 30 patients in the control group will only receive standard care, whilst waiting to receive actual treatment for their chronic pain. Intervention and control group will be compared on a number of outcome measures related to quality of life before using VR, during VR use, just after use and 4 months after final use. This explorative study is necessary to get first insights as a basis for a confirmative study.

DETAILED DESCRIPTION:
Rationale:

21,2% of the Dutch population is suffering from chronic low-back pain. 90% of these patients suffers from chronic low-back pain not attributable to a recognisable, specific pathology (non-specific low-back pain). 30-40% of all patients suffering from chronic pain visit their GP for treatment. Treatment includes mostly analgesics, in particular NSAIDs and opioids.

Adequate treatment of chronic pain is important as chronic pain negatively impacts, amongst others, quality of life, activities of daily living and feelings of helplessness. A systematic review by Bala et al. however shows that chronic pain treatment is often inadequate. Moreover, each different type of analgesic has its own associated side effects. NSAIDs increase the risk of cardiovascular and gastrointestinal complications. Common side effects of opioid analgesics include sedation, dizziness, nausea, vomiting, constipation, physical dependence, and even cases of hyperalgesia.

Recently, more attention has been given to psychological interventions for relieving chronic pain. A systematic review by Castelnuovo et al. shows the efficacy of a range of psychological interventions, including acceptance and commitment therapy (ACT), mindfulness-based interventions, hypnotherapy, eye movement and desensitization and reprocessing (EMDR) therapies and virtual reality based interventions. All of these psychological interventions focus on changing people's attitudes, feelings and behaviors on chronic pain, to improve their quality of life.

The first psychological intervention is the commonly used acceptance and commitment therapy (ACT). ACT is a cognitive behavioral therapy for treating chronic pain that uses exposure-based and experiential methods aiming at improving patients' abilities to cope with their chronic pain. Several systematic reviews indicate that ACT is effective in improving health outcomes of chronic pain patients. Mindfulness-based interventions seem to work as well for chronic pain relief. This set of interventions aims at learning strategies for pain awareness and acceptance. Furthermore, hypnotherapy is a mind-body based intervention that uses hypnoses to learn patients to cope with their pain. It focuses attention away from pain, thereby blocking its experience. Hypnotherapy seems effective in reducing pain experience. Then, eye movement desensitization and reprocessing (EMDR) is another psychotherapeutic approach in treating chronic pain. EMDR has already shown to be effective in treating posttraumatic stress disorder, and has recently as well been introduced as a treatment for chronic pain. Early research findings indicate EMDR to be effective in treating chronic pain.

Finally, one of the most recent fields of inquiry in treating chronic pain by means of psychological interventions is Virtual Reality. VR consists of a Head Mounted Device (HMD) and a sound system which immerses the user in a three-dimensional (3D) virtual world. There are multiple mechanisms behind the efficacy of VR in treating chronic pain. The most commonly studied mechanism is distraction. VR seems to be effective in reducing pain via distraction as it diverts attention away from pain. As both the VR application and the pain require attention and the brain has only limited attentional capacity, less attention is available for pain processing. In this manner, it reduces current feelings of pain, anxiety and stress. Though, the distraction mechanism only diverts attention away from pain shortly. To actually treat chronic pain by means of VR, it seems that other strategies, apart from distraction, are required.

Several studies aimed to find alternative mechanisms behind pain reduction by VR. The use of psychological interventions in VR, such as ACT or hypnosis, appears to be effective. Although the context of VR is different from traditional psychotherapy, the idea of how change occurs is not. Moreover, the immersiveness of VR provides opportunities to even better influence cognitions and emotions of patients suffering from chronic pain. Multiple virtual reality interventions have been designed with this knowledge in mind. A proof-of-concept study by Gromala et al., for example, looked into the application Virtual Meditative Walk (VMW). VNW focuses on mindfulness-based stress reduction via VR. The user study shows VNW's efficacy compared to non-VR interventions. Likewise, Guarino et al. proved that using virtual mindfulness therapy eight times over a period of a month is effective in chronic pain reduction. Therapeutic hypnosis has as well been tested in several case report studies. All conclude that virtual reality hypnosis seems to be effective in dealing with chronic pain.

The VR serious game Reducept is a novel psychological VR intervention for treating chronic pain. It incorporates several psychological therapies into one application: hypnotherapy, mindfulness, ACT and EMDR. Reducept has been made in co-creation with patients, researchers, psychologists and developers and can be installed and played on a VR goggles. It consists of an education module and three games.

* Education: Reducept provides its players with information about the biological mechanisms underlying chronic pain. Learning about chronic pain helps to cope with it in daily life.
* Control: Reducept's first game has been based on the mechanisms of hypnotherapy. The patient should shoot away painful stimuli in the nervous system. By visualizing their pain, they learn to control and cope with it.
* Relaxation: the second game within Reducept is a mindfulness-based intervention. It takes place in the spinal cord. Players should collect positive neurotransmitters and focus on their respiration rate.
* Processing: game three has been based on the mechanisms of ACT and EMDR. It asks players to recover negative patterns in the brain. Players have to switch attention between the pain and the game, helping them to decrease their experience of pain.

This study aims to gain a first understanding in the ability of the therapeutic VR intervention Reducept to treat chronic low-back pain. It will define a wide range of outcome measures, including quality of life indicators, pain, stress and anxiety measures and measures on ability to execute daily activities. What outcome measures does it affect? What outcome measures will be left unaffected? Moreover, tolerability, feasibility and acceptability of Reducept in relation to different patient characteristics (age, gender, Motivaction profiling) will be measured to understand which patients might benefit most from virtual reality based psychological interventions. The study focuses on patients with non-specific chronic low-back pain as this group represents a large part of all chronic pain patients. This explorative study is necessary as an input for future studies on the actual effects of therapeutic virtual reality interventions on quality of life of patients.

Objective:

To investigate whether a therapeutic virtual reality application can improve the quality of life of people suffering from non-specific chronic low-back pain, compared to a control condition.

Study design:

This explorative study uses a randomised controlled parallel design (1:1). Participants will be randomly assigned to either the control group or the intervention group. In the control group, participants are placed on the waiting list to receive the common treatment to handle their chronic pain. As they are placed on the waiting list, they will receive no therapeutic treatment yet (apart from the during intake prescribed physiotherapy and medication). Participants placed in the intervention group, who are also placed on the waiting list and only receive, when prescribed, physiotherapy and medication, will use the therapeutic virtual reality intervention meanwhile at home during a period of 28 days for at least ten minutes each day and in addition the education module at least during day 1 (which lasts 25 minutes). The randomisation is not blinded: both researchers and participants know which participants are part of the intervention and control group.

Study population:

Adult patients, males and females, suffering from daily non-specific chronic low-back pain are eligible for this study. Patients' pain should have last for at least three months. Patients should report a pain score of ≥4 during the intake questionnaires filled in before intake at the Rijnstate Pijncentrum.

Intervention (if applicable):

Participants will be randomly assigned to either the intervention group or the control group. Participants assigned to the intervention group will receive virtual reality glasses with the Reducept application. They are asked to use the therapeutic virtual reality intervention at home over a period of 28 days starting the day after collecting the virtual reality goggles. Participants are asked to use the therapeutic virtual reality intervention at least once a day for ten minutes. In addition, they should, on the first day, and preferably during more days, watch the whole education program which lasts 25 minutes. Participants can decide themselves to use the application more often. Participants assigned to the control group will receive no intervention, they are, just as the intervention group, placed on the waiting list to receive normal treatment.

Unfortunately, it is not possible to provide all patients with the opportunity to use the virtual reality application, as the design requires a control group that does not use it over the study period.

The investigators will study the possibility of continuing the virtual reality treatment for all participants want-ing to after finishing this study. At least they will be able to buy themselves the virtual reality glasses for using the therapeutic virtual reality.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

There is no risk involved in exposure to the therapeutic virtual reality application. Participants can leave the study at any time for any reason if they wish to do so without any consequences. As mentioned before, the burden for participants associated with this study is mainly related to measurements of endpoints, which will take approximately 30-45 minutes three times over a period of five months. The intervention group will spend at least ten minutes a day on the therapeutic virtual reality application and in addition on day 1 25 minutes.. As explained in the rationale, no or only minimal adverse effects from this intervention are expected.

ELIGIBILITY:
Inclusion Criteria:

1. Patient suffers from chronic non-specific low-back pain (LBP) not attributable to a recognisable, known speciﬁc pathology (e.g. infection, tumour, osteoporosis, lumbar spine fracture, structural deformity, inﬂammatory disorder, radicular syndrome, or cauda equina syndrome).
2. Patient reports a pain score related to chronic low-back pain ≥4.
3. Patient is placed on the waiting list to receive intervention and receives no treatment yet, apart from medication or physiotherapy.
4. At the day of recruitment, the estimated length of the waiting list for intervention is at least six weeks.
5. Patient did not receive any invasive treatment for his chronic non-specific low-back pain in the last year.
6. Patient is willing and able to comply with the trial protocol.
7. Patient is at least 18 years old on the day the oral informed consent will be given.
8. Patient can read and understand the Dutch language.

Exclusion Criteria:

1. Patient is included in another trial to evaluate new ways of treating pain.
2. Patients suffers from severe anxiety or depression (HADS≥16).
3. Patient has difficulties to handle virtual reality:

   1. Patient suffers from delirium or acute confusional state.
   2. Patient has (a history of) dementia, seizure, or epilepsy.
   3. Patient has severe hearing/visual impairment not corrected.
   4. The skin of the patient's head or face is not intact (for example head wounds, psoriasis, eczema).

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change in SF12: short form health survey | Day 0, day 28, day 148
  Measurement of changes in quality of life of patient before intervention, just after intervention period and 4 months after intervention period. SF12 measures via different scaled questions eight concepts: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. The first four items together form the physical health scale. The latter four items form the mental health scale. The higher the scores, the better the physical and mental health. Highest possible score: 56. Lowest possible score: 12.

SECONDARY OUTCOMES:
Change in positive health questionnaire | Day 0, day 28, day 148
  Measurement of changes in the positive health framework (a questionnaire and conversation tool for understanding health in a larger context) before intervention period, just after the intervention period and four months after the intervention period. Positive health consists out of 42 statements separated in 6 categories: bodily functioning, mental functioning, spiritual dimension, quality of life, social participation, daily functioning. Each question should be rated with a 0 (worst) to a 10 (best). The higher the scores, the better the quality of life.
Change in pain via numeric rating score | Day 0, day 28, day 148
  Measurement of changes in pain scores of patient before intervention period, just after intervention period and 4 months after intervention period. Pain scores are measured via a numeric rating score from 0 (no pain at all)-10 (worst pain ever). Questionnaire consists out of 4 questions, with a maximum score of 40.
Change in BPI: brief pain inventory, numeric rating score | Day 0, day 28, day 148
  Measurement of changes in pain inventory of patient before intervention period, just after intervention period and 4 months after intervention period. Questionnaire consists out of 7 questions to be answered with 0 (no obstruction) to 10 (full obstruction). A total of 70 points is the maximum score.
Change in PCS: Pain Catastrophizing Scale | Day 0, day 28, day 148
  Measurement of changes in pain catastrophizing of patient before intervention period, just after intervention period and 4 months after intervention period. Questionnaire consists out of 13 questions to be answered with 0 (not at all) to 4 (always). Questionnaire has 3 subscales (rumination, magnification, helplessness) and a total score of maximum 52.
Change in PCCL: Pain Coping and Cognition list | Day 0, day 28, day 148
  Measurement of changes in pain coping strategies (PCCL) of patient before intervention, just after intervention period and 4 months after intervention period. Questionnaire consists out of 42 questions to be answered with 0 (don't agree) to 5 (totally agree). 4 subscales: catastrophizing, pain coping, internal pain control, external pain control. Per subscale is the total sum calculated and divided by the number of questions. A score of 1-6 is assigned per subscale.
Change in HADS: Hospital Anxiety and Depression Scale | Day 0, day 28, day 148
  Measurement of changes in anxiety (HADS) of patient before intervention period, just after intervention period and 4 months after intervention period. Questionnaire consists out of 14 questions with answers ranging from 0 (often) to 3 (almost never). All questions are summed up to a total of 42 points.
Change in OLBPDQ: Oswestry Low Back Pain Disability Questionnaire | Day 0, day 28, day 148
  Measurement of changes in activities of daily life as a consequence of experienced pain of patient before intervention period, just after intervention period and 4 months after intervention period. Questionnaire consists out of 10 questions to be answered with 0 (no disability) to 6 (full disability). All questions are to be summed up to a total of 60 points.
Change in ADL: Activities of Daily Life | Day 0, day 28, day 148
  Measurement of changes in activities of daily life (ADL) of patient before intervention, just after intervention period and 4 months after intervention period. Questionnaire consists of 22 questions ranging from 0 (not at all) to 3 (easily autonomous). Maximum score is 63.
Change in pain questionnaire via numeric pain rating scale | Questionnaires will be filled in at the end of each intervention day during the intervention period of 28 days
  Changes in pain intensity during the intervention period measured via 4 questions on scales ranging from 0 (pain doesn't influence me) to 10 (pain hinders me a lot). And two visual analogue scales of 10 centimeters (I don't have pain at all - I am in full pain).
Medication use questionnaire | Questionnaires will be filled in at the end of each intervention day during the intervention period of 28 days
  Use of medication during the intervention period.

OTHER OUTCOMES:
Patient characteristics related to use of VR | Baseline (Questionnaire will be filled in once before the start of the intervention period.)
  Age, gender, education, employment, lifestyle, experience with technology - qualitative measures.
Feasibility of therapeutic virtual reality via semi structured interview | Semi-structured interviews with intervention group at intervention day 7,14 and 28
  Dosing and frequency of treatment, time of use, type of game. This will be monitored by the therapeutic virtual reality application itself.
  Reasons for use. Patient will be interviewed about issues during use of therapeutic virtual reality software/hardware.
Acceptability of therapeutic virtual reality via semi structured interview | Semi-structured interviews with intervention group at intervention day 7,14 and 28
  Patient will be interviewed about his or her opinion on therapeutic virtual reality hardware and software, patients' opinion on the effectiveness of therapeutic virtual reality, reasons to withdraw.
Tolerability of therapeutic virtual reality via semi structured interview | Semi-structured interviews with intervention group at intervention day 7,14 and 28
  Patient will be interviewed and asked about experienced adverse events, discomfort, inconveniences.

CONTACTS AND LOCATIONS:
Overall Officials: Harry van Goor, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Rijnstate, Velp, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Only upon asking.